CLINICAL TRIAL: NCT03409562
Title: Efficacy of Pain Neurophysiology Education in Combination With Motor Control Training for Patients With Unspecific Low Back Pain
Brief Title: Efficacy of Pain Neurophysiology Education in Combination With Motor Control Training for Unspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario Fundación Alcorcón (Other); FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Principal Investigator, Gustavo Plaza Manzano, Director, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI 17/108; 18/068-E (Other: CEIC Hospital Clínico San Carlos)
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Low Back Pain
Keywords: low back pain; pain neurophysiology education; motor control
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neurophysiology Education and motor control training (Experimental): This group will undergo two pain neurophysiology education sessions prior to motor control training.
  Interventions: Behavioral: motor control training; Behavioral: pain neurophysiology education
- motor control training alone (Active Comparator): This group will only perform motor control training.
  Interventions: Behavioral: motor control training

INTERVENTIONS:
Behavioral: motor control training — Exercises to strengthen the lumbar musculature and control the posture.
Behavioral: pain neurophysiology education — Educational sessions to improve patient's neurophysiology of pain knowledge.
  Other Names: pain neuroscience education
  Arms: Pain Neurophysiology Education and motor control training

SUMMARY:
The purpose of the present study is to evaluate whether the addition of two pain neurophysiology education sessions to motor control training may result in an improvement of the outcome measures of pain and disability, compared to motor control training alone.

DETAILED DESCRIPTION:
Sixty-two subjects with unspecific low-back pain were randomly recruited for the present study. The subjects were randomly allocated to a control group (which received only motor control training) and an intervention group (which underwent two pain neurophysiology education sessions prior to motor control training). Primary outcome measures were pain (measured with the Visual Analogical Scale) and disability (measured with the Oswestry Disability Index). Secondary outcome measures are kinesiophobia (Tampa Scale for Kinesiophobia), the global perceived effect (Global Perceived Effect Scale) and quality of life (SF-12). These will be measured before the intervention, at the end of the intervention, and 3 and 6 months after ending the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Unspecific low back pain for at least 3 months
* Patients must be knowledgeable in the language in which the educational sessions will be provided (Spanish)

Exclusion Criteria:

* Specific low back pain (e.g. infection, tumor, fracture, radiculopathy).
* Signs and symptoms of neuropathic pain or generalized chronic pain.
* History of lumbar or cervical spine surgery.
* Pregnancy.
* Concomitant pathologies that impede the performance of exercises.
* Psychiatric treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Change in pain at different time points | Assessed before the intervention, at the end of the 4-week motor control intervention and 3 and 6 months after the end of the intervention
  Visual Analogic Scale
Change in disability at different time points | Assessed before the intervention, at the end of the 4-week motor control intervention and 3 and 6 months after the end of the intervention
  Oswestry Disability Index

SECONDARY OUTCOMES:
Change in kinesiophobia at different time points | Assessed before the intervention, at the end of the 4-week intervention and 3 and 6 months after the end of the intervention
  Tampa Scale of Kinesiophobia
Change in Global Perceived Effect at different time points | Assessed before the intervention, at the end of the 4-week motor control intervention and 3 and 6 months after the end of the intervention
  Global Perceived Effect Scale
Change in quality of life at different time points | Assessed before the intervention, at the end of the 4-week motor control intervention and 3 and 6 months after the end of the intervention
  SF-12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plaza-Manzano, Ph.D, Study Director — Universidad Complutense de Madrid
Locations (2):
- Spain (2):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Clínico San Carlos, Madrid